CLINICAL TRIAL: NCT06586970
Title: Tailored Occupational Therapy and Registered Dietitian Services for Home-Delivered Meal Clients: A Randomized Controlled Trial
Brief Title: Occupational Therapy and Registered Dietitian Services to Reduce Fall Risk Among Home Delivered Meal Clients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: LifeCare Alliance (Unknown)
Responsible Party: Principal Investigator, Lisa Juckett, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 90INNU0044-01-00; 90INNU0044-01-00 (Other Grant/Funding Number: Administration for Community Living)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Diet, Food and Nutrition; Accidental Falls; Cardiovascular Diseases; Diabetes; Debility; Frailty; Functional Disability
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Frailty | interventions — Meals

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Meals only (No Intervention): ARM 1: Meals only. Participants randomized to receive "meals only" will receive 7-14 frozen meals, delivered 1x/week, for 3-months. Participants will be provided with a menu of 42 meal options and instructions for how to select their meals and change weekly meal selections (if desired). Participants in this arm will also receive nutrition education and fall prevention handouts. Nutrition education handouts will indicate which of LifeCare Alliance's meals are considered to be "heart healthy" as well as "diabetic-friendly." Participants will have the autonomy to select their own meals according to their preferences and their ability to self-manage their own health conditions (e.g., diabetes, cardiovascular disease). Fall prevention education handouts will provide guidance on how to reduce fall risk at home and modify the home environment to eliminate fall hazards.
- Arm 2: Meals + RD services (Active Comparator): ARM 2: Meals + registered dietitian services. Participants randomized to receive "meals + RD only" will receive 7-14 frozen meals, delivered 1x/week, for 3-months. In addition to receiving nutrition education and fall prevention handouts, participants in this arm will have a telephone-based nutrition assessment completed by one of LifeCare Alliance's registered dietitians who will assign participants a nutrition diagnosis (e.g., overconsumption of carbohydrates) within 60 days of study enrollment.
  Interventions: Behavioral: Meals + RD services
- Meals + OT services (Active Comparator): ARM 3: Meals + occupational therapy services. Participants randomized to this arm will receive 7-14 frozen meals, delivered 1x/week, for 3-months and be able to make weekly meal selections from LifeCare Alliance's full list of 40 meals. In addition to receiving nutrition education and fall prevention handouts, participants in this arm will be contacted (within 30 days of study enrollment) by one of Lifecare Alliance's occupational therapists to complete a phone screen to determine each participant's occupational therapy needs (e.g., home safety/fall risk hazards, need for durable medical equipment).
  Interventions: Behavioral: Meals + OT services
- Arm 4: Meals + RD + OT services (Active Comparator): ARM 4: Meals + registered dietitian services + occupational therapy services. Participants in this arm will receive 7-14 frozen meals, delivered 1x/week, for 3-months as well as the same nutrition education and fall prevention handouts as provided in Arms 1-3. Additionally, participants will receive the combination of dietitian and OT services as provided in Arms 2 and 3 and have the same autonomy to make their own weekly meal selections from a curated list provided by the dietitian.
  Interventions: Behavioral: Meals + RD + OT services

INTERVENTIONS:
Behavioral: Meals + RD services — Registered dietitians (RD) will provide tailored dietitian counseling and nutrition education
  Arms: Arm 2: Meals + RD services
Behavioral: Meals + OT services — Occupational therapists (OT) will provide tailored home safety recommendations and fall prevention education/strategies
  Arms: Meals + OT services
Behavioral: Meals + RD + OT services — A combination of tailored registered dietitian and occupational therapy services will be provided
  Arms: Arm 4: Meals + RD + OT services

SUMMARY:
The purpose of this study is to determine which of the following four service models is most effective for reducing fall risk among home-delivered meal clients: (1) meals alone, (2) meals + registered dietitian services, (3) meals + occupational therapy services, (4) meals + registered dietitian + occupational therapy services.

DETAILED DESCRIPTION:
Home delivered meal programs provide essential health and nutritional support to community-dwelling older adults in the United States. Without this support, nearly three million older adults would be at even greater risk for malnourishment and subsequent health decline, leading to potential hospitalizations and nursing home placements. Despite the reported value of home delivered meals, the increasingly complex health needs of the older adult population warrant new, innovative approaches that enhance home-delivered meal services. In our prior work, we identified that the majority of home delivered meal clients are at high risk for malnutrition, increasing clients' risk of falling and warranting the need for registered dietitian services to attenuate health decline. Additionally, our other work has identified that 80% of home delivered meal clients are at elevated risk for falling,6 and over 40% have experienced a fall in the past year. The high prevalence of fall risk factors among home delivered clients suggests that additional services - such as occupational therapy - are also needed to optimize clients' ability to safely remain living in their own homes and communities. In response to home delivered meal clients' need for more enhanced and specialized services, the present study will test four different service models to determine which model is most effective for reducing fall-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to receive meals according to LifeCare Alliance's standard in-take criteria (Over the age of 60; unable to safely and independently leave the home; does not have access to a caregiver who can prepare meals)
* Has a working freezer to store between 7-14 frozen meals/week
* Has a working microwave or oven to reheat meals
* Lives within LifeCare Alliance's 5-county service area

Exclusion Criteria:

* Individuals already receiving home-delivered meals from LifeCare Alliance or other meal agency (within the past 40 days)
* Individuals residing in residential care or a skilled nursing facility
* Individuals whose dietary restrictions prohibit them from eating meals from LifeCare Alliance's frozen meal selection
* Individuals at home on hospice care
* Unable to independently answer LifeCare Alliance's in-take questions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Falls Efficacy Scale | Baseline; 3-months; 6-months
  Questionnaire to assess concerns with falling during routine activities of daily living; scores range from 7-28 points with lower scores indicating a lower concern with falling

SECONDARY OUTCOMES:
Mini Nutritional Assessment-Short Form | Baseline; 3-months; 6-months
  Questionnaire to assess risk of malnutrition; scores range from 0-14 points with lower scores indicating a lower risk of malnutrition
Dietary intake | Baseline; 3-months; 6-months
  Four items drawn from the Summary of Diabetes Self-Care Activities questionnaire to assess quality of foods consumed; scores range from 0-28 with higher scores indicating consumption of higher quality foods
EQ-5D-5L | Baseline; 3-months; 6-months
  Five domain measure to assess quality of life in the areas of mobility, self-care, usual activities, pain/discomfort and anxiety/depression; scores range from 5 to 25 points with lower scores indicating better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- LifeCare Alliance, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is not required by our funder and is not of interest to our partner agency who is leading the provision of the interventions being tested